CLINICAL TRIAL: NCT03637270
Title: Incorporating Supplementary Protein Into Rehabilitative Exercise (INSPIRE Trial) for Patients With Chronic Stroke
Brief Title: Protein Supplementation for Chronic Stroke Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Principal Investigator, Yen-Nung Lin, Director of Department of Rehabilitation, WanFang Hospital, Taipei Medical University WanFang Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 107-2320-B-038 -016
Record Dates: First submitted 2018-08-15; First posted 2018-08-17 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Chronic Stroke
MeSH Terms: interventions — Dietary Supplements; Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRO group (Experimental): Participants in PRO group receive dietary supplementation with protein-rich supplements immediately before and after each exercise training session. The interventions include 30 training sessions.
  Interventions: Dietary Supplement: Dietary supplementation; Other: Exercise training
- CHO group (Active Comparator): Participants in CHO group receive dietary supplementation with carbohydrate-rich supplements immediately before and after each exercise training session. The interventions include 30 training sessions.
  Interventions: Dietary Supplement: Dietary supplementation; Other: Exercise training

INTERVENTIONS:
Dietary Supplement: Dietary supplementation — Before and after each exercise session, the research assistant will give subjects protein supplement or carbohydrate supplement according to the treatment assignment and ask them to drink it down right away.
Other: Exercise training — Including aerobic cycling training and progressive resisted exercise

SUMMARY:
Stroke patients usually have difficulties with moving and are venerable to secondary problems such as sarcopenia and strength loss. These problems may accelerate the disability process during aging. It is well known that exercise helps to maintain or promote human fitness. This study is conducted to explore the beneficial effects of exercise and protein supplement on fitness and body composition among patients with chronic stroke.

DETAILED DESCRIPTION:
This is a multicenter randomized control trial. Participants will be recruited from 4 teaching hospitals in Taipei. Participants are randomly assigned to 2 groups:

1. protein supplementation + exercise (PRO group);
2. carbohydrate supplementation + exercise (CHO group);

The 1-hour exercise intervention includes aerobic cycling exercise followed by progressive resisted exercise with TheraBand. PRO group receives PS immediately before and after the exercise while the CHO group receive sham product (the same calories with no protein). The Interventions are arranged 3 sessions a week for 10 weeks. The outcome measurements are performed at 0-week, 10-week, and 20-week.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic stroke>6months
2. Age : 20-75 y
3. Able to walk independently over 10 mins (with or without orthosis)
4. Able to use stationary bike

Exclusion Criteria:

1. Physiological condition not stable, cognitive dysfunction, not able to coordinate with examine or treatments.
2. Not able to exercise due to severe cardiopulmonary dysfunction
3. Malnutrition (MNA<11)
4. Severe obesity (BMI>35)
5. Renal insufficiency
6. Unable to tolerate our cardiopulmonary exercise test (CPET) (eg, too short stature to fit the machine, leg spasticity is too strong to peddle the cycling, unable to maintain 50 rpm at the beginning of CPET, indications for early termination of CPET based on the American College of Sport Medicine suggestions)

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2018-12-19 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-03 (Actual)

PRIMARY OUTCOMES:
Cardiopulmonary capacity | 10 weeks
  VO2-peak. Oxygen consumption (VO2- peak) were measured during our cardiopulmonary test (with a ramped stationary biking and a gas analyzer). The workload was increased at a ramp rate of 5-10 W/min. A cadence at 50~70 rpm was to be maintained.

SECONDARY OUTCOMES:
Total body lean and fat mass | 20 weeks
  measured by dual energy X-ray absorptiometry
Timed up and go (TUG) | 20 weeks
  measures the mixed capacity of balance and walking
Burg Balance Test | 20 weeks
  measures the balance
CardioPulmonary Exercise Test | 20 weeks
  measures cardiopulmonary fitness
6 minutes walk test | 20 weeks
  measures the walking endurance
Physical performance (short physical performance battery) | 20 weeks
  measured by clinical evaluation
Physical performance (modified physical performance test) | 20 weeks
  measured by clinical evaluation
Maximal isometric voluntary contraction | 20 weeks
  measured by clinical evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Yen-Nung Lin, MD, MS, Principal Investigator — Department of Physical Medicine and Rehabilitation, Wan-Fang Hospital, Taipei Medical Univerisity
Locations (4):
- Taiwan (4):
  - Department of rehabilitation, Shuang-Ho Hospital, New Taipei City
  - Department of rehabilitation, Taipei Tzu-Chi Hospital, New Taipei City
  - Department of rehabilitation, Taipei Medical University Hospital, Taipei
  - Department of rehabilitation, WanFang Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No